CLINICAL TRIAL: NCT00010712
Title: Effects of Black Cohosh on Menopausal Hot Flashes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: P50AT000090-01P3 (NIH); P50AT000090-01 (NIH); NCT00009386 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Postmenopause; Hot Flashes; Osteoporosis, Postmenopausal
Keywords: Menopause; Hot Flashes; Osteoporosis; Postmenopausal
MeSH Terms: conditions — Hot Flashes; Osteoporosis, Postmenopausal; Osteoporosis | interventions — black cohosh root extract

INTERVENTIONS:
Drug: Black Cohosh

SUMMARY:
This study will assess whether treatment with black cohosh is effective in reducing the frequency and intensity of menopausal hot flashes. In addition, this study will determine whether or not black cohosh reduces the frequency of other menopausal symptoms and improves quality of life.

DETAILED DESCRIPTION:
Most American women will spend the last third of their lives post-menopause. During this time, chronically low levels of steroidal estrogens may lead to a number of short and long-term medical sequelae such as hot flashes, vaginal dryness, heart disease, and osteoporosis. While some physicians believe that demonstrated beneficial effects of estrogen, particularly on the cardiovascular and skeletal systems, warrant the taking of hormone therapy from menopause on, many women choose not to take estrogen replacement therapy (ERT) and are increasingly exploring alternative approaches to ERT.

For centuries, black cohosh (Cimicifuga racemosa) has been used worldwide for women's health. Despite its long-standing use, studies of black cohosh have yielded conflicting data, in part because of lack in study design rigor and the short duration of studies to date. The primary aim of this study is to correct past shortcomings in study design to determine whether treatment with black cohosh is effective in treating menopausal symptoms.

Participants in this study will be given black cohosh for a 12-month period. Potential mechanisms of action of black cohosh will be examined by quantifying the levels of sex hormones, including estradiol, estrone, FSH, and LH. Because black cohosh may act as an estrogenic agent, the effect on endometrium will be evaluated by sonogram and by monitoring the incidence of adverse events and compliance with the study.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the New York Metro Area
* Postmenopausal
* Weight within 90% to 120% of ideal body weight

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Fredi Kronenberg, Principal Investigator — Columbia University
Locations (1):
- Columbia University Rosenthal Center for CAM, New York, New York, United States